CLINICAL TRIAL: NCT00175721
Title: Randomized Controlled Trial Comparing Current Care in Multiple Clinics Vs Care in a Novel Cardiac, Diabetes & Kidney Care Clinic
Brief Title: Trial Comparing Care in Multiple Clinics Versus Care in a Cardiac, Diabetes and Kidney Care Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H04-50008
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Kidney Diseases; Heart Diseases; Diabetes Mellitus
Keywords: Combined Clinic; Chronic Kidney Disease; Diabetes
MeSH Terms: conditions — Kidney Diseases; Heart Diseases; Diabetes Mellitus; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: The Combined Cardiac Kidney Diabetes Care Clinic — See Detailed Description.

SUMMARY:
The purpose of this study is to assess the benefits of a combined cardiac, kidney, and diabetes clinic versus multiple clinics.

Hypothesis: Attendance at multiple clinics by one individual patient has multiple problems which may be overcome by the introduction of a combined care clinic.

DETAILED DESCRIPTION:
This is a randomized control trial to compare health care resource utilization, and achievement of stated targets of therapy (BP, Hgb, glucose control, use of preventive medications) as well as patient and health care team satisfaction, and longer term patient outcomes in patients with kidney disease who have either or both diabetes and heart disease, and currently attend either a diabetic or heart function clinic (or both) in addition to a kidney care clinic. In addition, we will also establish and refine the specialized cross-disciplinary care model, within a framework in Vancouver, and evaluate its functioning from the perspectives of allied health and medical professionals.

This is a systematic evaluation of health care delivery methods to a complex group of patients, which will serve as a nidus for ongoing research in both health outcomes research, and biomedical research.

The creation of this multifaceted clinic in an organized manner would permit evaluation of all of the components of it, and also demonstrate the importance of collaboration between disciplines and between public health care initiatives and industry partners, who would fund this clinic infrastructure and research components in the initial phase.

ELIGIBILITY:
Inclusion Criteria:

* All patients currently attending or who would be eligible to attend 2 or more of the following clinics: cardiac, diabetic or kidney

Exclusion Criteria:

* Those patients currently attending the diabetic, cardiac or kidney clinics who do not have more than one condition (i.e. who have only one of the diagnoses) or who refuse to sign informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Health care utilization and patient/provider satisfaction (5 years) | 5 years

SECONDARY OUTCOMES:
Patient outcomes (5 years) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Adeera Levin, MD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada